CLINICAL TRIAL: NCT01949792
Title: An Open-label Single- and Multiple-dose Trial Investigating the Pharmacokinetics and Pharmacodynamics of rFVIIa Following i.v. Administration of One Dose of 270 Microg/kg and Three Doses of 90 Microg/kg in Patients With Haemophilia A or B With or Without Inhibitors
Brief Title: A Trial Investigating the Pharmacokinetics and Pharmacodynamics of rFVIIa in Patients With Haemophilia A or B With or Without Inhibitors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: NN7777-4086; 2013-000040-26 (EudraCT Number); U1111-1138-2521 (Other: WHO)
Record Dates: First submitted 2013-09-13; First posted 2013-09-25 (Estimated); Last update posted 2014-11-14 (Estimated); Status verified 2014-11

CONDITIONS: Congenital Bleeding Disorder; Haemophilia A; Haemophilia A With Inhibitors; Haemophilia B; Haemophilia B With Inhibitors
MeSH Terms: conditions — Hemophilia A; Hemophilia B | interventions — Factor VII

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 270 microg/kg rFVIIa (Active Comparator): Each subject will receive one single injection of 270 microg/kg and three injections of 90 microg/kg rFVIIa (one injection every 3 hours) in a randomised order. The two administration days will be separated by a wash-out period of at least 48 hours
  Interventions: Drug: eptacog alfa (activated)
- 3x90 microg/kg rFVIIa (Active Comparator): Each subject will receive one single injection of 270 microg/kg and three injections of 90 microg/kg rFVIIa (one injection every 3 hours) in a randomised order. The two administration days will be separated by a wash-out period of at least 48 hours
  Interventions: Drug: eptacog alfa (activated)

INTERVENTIONS:
Drug: eptacog alfa (activated) — Subject will receive a single injection (i.v.) of 270 microg/kg rFVIIa (NovoSeven®)
  Arms: 270 microg/kg rFVIIa
Drug: eptacog alfa (activated) — Subject will receive 3 injections (i.v.) of 90 microg/kg rFVIIa (NovoSeven®) over a 6 hour period (each injection will be separated by 3 hours)
  Arms: 3x90 microg/kg rFVIIa

SUMMARY:
This trial is conducted in Europe. The aim of the trial is to investigate the pharmacokinetics (the exposure of the trial drug in the body) and pharmacodynamics (the effect of the investigated drug on the body) of rFVIIa (activated coagulation factor VII) following one single injection of 270 microg/kg compared to three injections of 90 microg/kg rFVIIa in patients with haemophilia.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent obtained before any trial-related activities. Trial-related activities are any procedures that are carried out as part of the trial, including activities to determine suitability for the trial
* Male patients with confirmed diagnosis of severe congenital haemophilia A or B (higher than 1% FVIII or FIX) with or without inhibitors to coagulation factors VIII or IX, based on medical records

Exclusion Criteria:

* Congenital or acquired coagulation disorder other than congenital haemophilia A or B
* Any clinical signs or known history of arterial thrombotic events or previous deep vein thrombosis or pulmonary embolism (as defined by available medical records)
* Use of any anticoagulant (e.g. un-fractionated or low molecular weight heparin, vitamin-K antagonists, direct thrombin inhibitors or factor Xa inhibitors)
* Bleeding prophylactic treatment or FVIII or FIX immune tolerance induction (ITI) treatment during the trial period

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2013-09; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Thromboelastography (TEG) parameter Maximum Thrombosis Generation (MTG;'maximum velocity') | 10 minutes post-dose for 270 microg/kg and 10 minutes after the first injection of 90 microg/kg

SECONDARY OUTCOMES:
TEG parameters r-time, MTG, alpha angle, and maximum amplitude (MA) | Prior to and 24 hours following the administrtion of 270 microg/kg and each of the 3 administrations of 90 microg/kg

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (1):
- Madrid, Spain

REFERENCES:
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com